CLINICAL TRIAL: NCT06710301
Title: Study of the Cortical Correlates of Spatial Navigation Skills in an Immersive Virtual Reality Environment
Brief Title: Cortical Correlates of Spatial Navigation Skills in an Immersive Virtual Reality Environment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Eugenio Medea (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1111
Record Dates: First submitted 2024-11-25; First posted 2024-11-29 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Cerebral Palsy (CP)
Keywords: Navigation skills; EEG; Virtual Reality; Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Navigation task (Experimental): Administration of the navigation task in an immersive virtual reality environment with recording of the EEG signal
  Interventions: Other: Preliminary assessment; Other: Navigation task with EEG recording

INTERVENTIONS:
Other: Preliminary assessment — Evaluation of the cognitive level through the Raven test and of spatial navigation skills through the Corsi test and the maze sub-test of the WISC-III.
Other: Navigation task with EEG recording — Administration of the navigation task in an immersive virtual reality environment and EEG signal recording. The participant will wear virtual reality viewers and EEG cap. The task consists in moving and orienting themselves inside a five-way maze in order to reach a treasure. The participant will be asked to carry out 30 trials lasting a maximum of 120s each.

SUMMARY:
The goal of this study is to investigate the neural mechanisms that undergoes spatial navigation skills in children/adolescents aged between 8 and 17 years. These skills play an important role in daily life, as they allow us to orient ourselves in familiar and unfamiliar environments, locate objects, interact with them and memorize their position. Navigation abilities vary widely between individuals, change with age and might be affected by diseases, such as the cerebral palsy (CP). Previous studies have, in fact, demonstrated differences in the learning and adaptation methods of spatial navigation skills in children affected by CP compared to typically developing (TD) peers. Through the use of the electroencephalogram (EEG) we want to shed light on the mechanisms that govern this ability with the aim of:

1. better characterize spatial navigation skills in children/adolescents, both TD and affected by CP;
2. investigate the origin of the differences found between the spatial navigation skills of TD children and those affected by CP, improving knowledge of the pathology and thus allowing, in the future, to identify more adequate rehabilitation interventions.

ELIGIBILITY:
Inclusion Criteria:

* typically developing subjects aged between 8 and 17 years;
* subjects with CP aged between 8 and 17 years;

Exclusion Criteria:

* subjects aged under 8 or over 17 years;
* subjects with epileptic problems;
* subjects with poor head control;
* subjects with visual problems that can not be corrected with prescription lens;

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2024-11-14 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Power Spectral Density (PSD) | Once
  Differences in power values between TD and CP subjects
Navigation performance | Once
  Navigation performance based on the following parameters: number of routes visited in each trial; total length of the path for each trial; error between distance traveled and ideal distance for each trial (identified as the minimum distance to reach the treasure from the starting point); angle of rotation of the viewer in each trial; duration of each trial.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - IRCCS Scientific Institute E. Medea, Bosisio Parini, LC
  - IRCCS Scientific Institute E. Medea, Conegliano, TV

IPD SHARING:
Plan to Share IPD: No